CLINICAL TRIAL: NCT06059300
Title: Digital Breast Tomosynthesis for the Dutch National Breast Cancer Screening Program
Acronym: STREAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); UMC Utrecht (Other); LRCB Dutch Expert Centre for Screening (Unknown); Dutch Breast Cancer Association (Unknown); University of Sydney (Other); Hologic B.V. (Unknown); Volpara Health Technologies Ltd (Unknown); Lunit Inc. (Industry); Screenpoint Medical BV (Unknown); Sectra Benelux (Unknown); iCAD (Unknown); Dutch Foundation of Population Screening (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 114374; 13710 (Other Grant/Funding Number: KWF); 5550402130002 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2023-07-17; First posted 2023-09-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Screening
Keywords: Digital breast tomosynthesis; Acceptability; Reading strategy; Artificial intelligence; Cost-effectiveness; Recall rate; Detection rate; Advanced cancer detection rate; Interval cancer rate
MeSH Terms: interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): 18200 participants who will be screened with tomosynthesis instead of digital mammography. All participants will be asked to participate in the study for 2 screening rounds. The number of participants for the second round will be less, due to drop-outs.
  Interventions: Diagnostic Test: Digital Breast Tomosynthesis

INTERVENTIONS:
Diagnostic Test: Digital Breast Tomosynthesis — Screening with Digital Breast Tomosynthesis instead of Digital Mammography, for two screening rounds

SUMMARY:
Digital breast tomosynthesis (DBT) creates a digital pseudo- three-dimensional image of the breast similar to mammography. This gives the screening radiologist more information about a possible abnormality. As a result, breast cancer can be found earlier, but more women might need to be recalled.

In the STREAM study, the aim is to identify the impact of DBT on the screen-detected cancer and recall rates, and on interval and advanced cancer rates in 18,200 women after two rounds of screening. For comparison, a control group of about 86,400 women will be selected from the database of the national screening program. Women, screening radiographers, and screening radiologists will be asked whether they find this new screening technique acceptable. Furthermore, the optimal strategy for screening radiologists to read the DBT images will be identified and the cost-effectiveness of screening with DBT will be determined. The images and data will be stored in a database for future research.

Expected outcome:

As a result of this project, the researchers will have shown if breast cancer screening with DBT in the Netherlands should be implemented or not. It will also be demonstrated, were it to be introduced, how it should be implemented, having addressed all the remaining questions, and having found the optimal DBT workflow specifically for a high-volume population-based screening program.

DETAILED DESCRIPTION:
In the last decade, several large-scale European studies have shown that digital breast tomosynthesis (DBT) increases the detection rate from ~6 to ~9 cancers per 1000 women screened, while the recall rate approaches 3.5% to 4%, independent of the initial recall rate. In the Dutch screening setting with digital mammography (DM), the recall rate is only 2.4%. Therefore, introducing DBT in the Netherlands will likely generate an increase in false positives, but the magnitude of this increase is unknown.

Furthermore, the ~50x increase in the number of images resulting from a DBT exam compared to a DM exam doubles the reading time. For DBT screening in the Netherlands to be feasible from the economic and human resources point of view, the interpretation of these cases must be accelerated, to result in an average reading time comparable to that of reviewing DM exams.

The aim of this project is to make the replacement of DM with DBT in the Dutch National Breast Cancer Screening Program feasible and sustainable, by ensuring its acceptability by the various stakeholders, optimizing the acquisition and reading strategy, determining its expected impact on the national recall rate, and determining its cost-effectiveness. In addition, completion of this project will result in the creation of a DBT-based screening database available for future research.

Work Package (WP) 1 will involve the introduction of DBT in 6 of the 71 screening units in the country to screen 18,200 women for two screening rounds. This study is powered to detect a combined one-third reduction in the interval and advanced cancer rates with DBT screening as the primary endpoint. In addition, as secondary endpoints, the Dutch DBT-based screening recall rates will be determined for the first and second rounds of DBT screening. A contemporary control group of about 86,400 women screened with DM will be selected from the screening database (ScreenIT) of the national screening program. This control group will be selected to reflect the distribution of urban and rural areas as well as the mixture of mobile and fixed units of the screening units selected for the intervention group. In addition, the attendees, and the screening radiographers and radiologists will be surveyed to identify any barriers that limit acceptability of this new modality. Finally, WP1 will also involve the creation of a DBT-based screening database for further research.

In WP2, the optimal DBT reading strategy to be used in the Dutch screening program to minimize the increase in reading time with DBT, will be identified. For this, retrospective observer studies will be performed, using the images from WP1, to test eight different acquisition and reading strategies, some involving the use of cutting-edge artificial intelligence computer systems. These strategies have been shown in initial studies, many performed by the sponsor, to result in a significant reduction in reading time, with no or minimal loss in performance. Once the optimal reading strategies is identified, it will be used to interpret the entire second round of DBT screening acquired in WP1 at the screening reading units retrospectively. In this way, its actual performance and impact on reading time in the real screening environment will be determined.

Finally, in WP3, the results from the other two WPs will be used to model the entire DBT screening program and therefore predict the long-term outcomes and cost-effectiveness of this new screening program. The only method possible to estimate the impact of screening on long-term effects, such as breast cancer mortality and morbidity, as well as cost-effectiveness, is the use of modelling. Therefore, the well-validated MISCAN model will be used, with the data and results gathered, to estimate the long-term impact of DBT screening.

As a result of this project, if successful, breast cancer screening with DBT will be ready for nationwide implementation, having addressed all the country-specific questions and having optimized the DBT workflow specifically for a high-volume population-based screening program.

ELIGIBILITY:
Inclusion Criteria:

* Women who are invited to participate to the Dutch Breast Cancer Screening program in the age group 50-72 years..

Exclusion Criteria:

* Disabled women
* Women who are wheelchair bound

Ages: 50 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18200 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
The effect of DBT screening on breast cancers diagnosed at an advanced stage at screening or in between rounds of screening. (detection rate of stage II+ cancers per 1000 screens and interval cancer rate per 1000 screens) | 5 years
  The outcome will be compared to the control group (DM)

SECONDARY OUTCOMES:
Attendance rate (percentage out of all women invited) | 5 years
  The outcome will be calculated for the intervention group (DBT) and the control group (DM):
Recall (percentage out of all women screened) | 5 years
  The outcome will be calculated for the intervention group (DBT) and the control group (DM):
Cancer detection rate for breast cancer, both invasive and in situ, overall and for cancers stage II or higher (stage II+; per 1000 screened) | 5 years
  The outcome will be calculated for the intervention group (DBT) and the control group (DM):
Positive predictive value for recall (percentage of cancers detected among recalled women) | 5 years
  The outcome will be calculated for the intervention group (DBT) and the control group (DM):
Interval cancer rates (breast cancer detected clinically in the first, second, or third year after a negative screening examination. | 5 years
  The outcome will be calculated for the intervention group (DBT) and the control group (DM):

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Broeders, Prof., Principal Investigator — Radboud University Medical Center; Ioannis Sechopoulos, Prof., Principal Investigator — Radboud University Medical Center; Nicolien van Ravesteyn, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Bevolkingsonderzoek Nederland, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The following end products will be made available for further research and verification:
  * Summary outcomes of the screening
  * Methods used during the study such as, but not limited to, data extraction algorithms, statistical analysis, and cost effectiveness
Supporting Information: Study Protocol, ICF
Time Frame: For the duration of the study

REFERENCES:
- See also: STREAM website — https://www.radboudumc.nl/lopende-onderzoeken/stream